CLINICAL TRIAL: NCT05036551
Title: Relationship Between Kinesiophobia, Pain, Functional Status and Self-Efficacy in Patients With Knee Osteoarthrıtıs
Brief Title: Kinesiophobia, Pain, Functional Status and Self-Efficacy in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Research assistant, Hacettepe University
Other Study IDs: HU-FTR-NK-01
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Kinesiophobia; Pain; Functional Status; Self Efficacy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Kinesiophobia; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 2 Knee osteoarthritis: The Visual Analogue Scale (VAS) was used to determine the severity of the pain. Tampa Scale for Kinesiophobia (TSK) was used to evaluate kinesiophobia. The functional state was evaluated using The Western Ontario and McMaster Universities Arthritis Index (WOMAC). The Arthritis Self Efficacy Scale was used to determine self efficacy perception.
  Interventions: Diagnostic Test: Kellgren Lawrence classification
- Stage 3 Knee osteoarthritis: The Visual Analogue Scale (VAS) was used to determine the severity of the pain. Tampa Scale for Kinesiophobia (TSK) was used to evaluate kinesiophobia. The functional state was evaluated using The Western Ontario and McMaster Universities Arthritis Index (WOMAC). The Arthritis Self Efficacy Scale was used to determine self efficacy perception.
  Interventions: Diagnostic Test: Kellgren Lawrence classification

INTERVENTIONS:
Diagnostic Test: Kellgren Lawrence classification — The Kellgren Lawrence classification was used in the radiological evaluation. It is a classification method used in the staging of knee osteoarthritis. Five stages were defined according to the anteroposterior X-ray.(Stage 0-5)

SUMMARY:
Objective: The aim of this study is to examine the relationship between kinesiophobia, pain, functional status and self efficacy in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Material and Methods: The study was performed on 72 individuals diagnosed with Stage 2 and Stage 3 knee osteoarthritis according to the Kellgren Lawrence classification. The Tampa Scale for Kinesiophobia (TSK) was used to evaluate kinesiophobia, and the Visual Analogue Scale (VAS) was used to assess pain. The Western Ontario and McMaster Universities Arthritis Index (WOMAC) was used to asses the functional status. Self efficacy was assessed using the Arthritis Self Efficacy Scale (ASES).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-85 and diagnosed with stage 2-3 bilateral knee osteoarthritis according to Kellgren Lawrence classification.

Exclusion Criteria:

* With a history of lower extremity surgery and a major trauma, orthopedic knee injuries such as tendinopathy, bursitis, ligament and meniscus injuries, a neurological or cardiopulmonary disease that may affect the evaluations, and any other joint in the lower limb that may cause reflected pain in the knee, individuals who had inflammatory rheumatic disease such as gout, rheumatoid arthritis, have participated in physical therapy and rehabilitation program in the last 6 months and who have been given knee injections

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | After the participants were examined, evaluations were made before starting the physical therapy program.
  Pain assessment, between 0-10 points. Low score low pain
Tampa Scale for Kinesiophobia | After the participants were examined, evaluations were made before starting the physical therapy program.
  Kinesiophobia assessment, between 17-68 points. Low score low kinesiophobia.
The Western Ontario and McMaster Universities Arthritis Index | After the participants were examined, evaluations were made before starting the physical therapy program.
  Functional state assessment, between 0-96 points. Low score good functional status.
Arthritis Self Efficacy Scale | After the participants were examined, evaluations were made before starting the physical therapy program.
  Self Efficacy assessment, between 20-100 points. Low score low self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hacettepe Üniversity, Intitue, Study Director — Hacettepe University Health Sciences Institute; Nurhayat Korkmaz, PhDstudent, Principal Investigator — Hacettepe University Health Sciences Institute
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)